CLINICAL TRIAL: NCT01956331
Title: Comprehensive Geriatric Assessment and Complications Following Lung Resection for Lung Cancer - A Prospective Observational Study in Elderly Patients With Non-small Cells Lung Cancer
Brief Title: Comprehensive Geriatric Assessment and Complications Following Lung Resection for Lung Cancer
Acronym: OPERAGE
Status: Completed | Type: Observational
Sponsor: Groupe Francais De Pneumo-Cancerologie (Other)
Responsible Party: Sponsor
Other Study IDs: GFPC 08-05
Record Dates: First submitted 2013-09-29; First posted 2013-10-08 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: NSC lung Cancer,Elderly patients,post operative,
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
schema : Prospective prognostic study The main objective is to study the value of the Comprehensive Geriatric Assessment in predicting the risk of post operative complications after lung resection for cancer.

DETAILED DESCRIPTION:
Primary outcome :

Post-operative morbidity at 30-day :

Post operative complications occurred during 30 days post surgery, evaluated with CTCAE V3.0, and Complications grade 2.3.4 will be analyzed from day 1, at day 20 up to day 30.

Evaluation :

Pre operative : Day -30 to Day 0, Post operative : Day 10, Day 30, Day 90, Day 360.

Secondary outcome :

Post-operative mortality, Length of post operative hospital stay, Length of intensive care unit stay, QOL assessment, One year survival.

ELIGIBILITY:
Inclusion Criteria:

* Patient 70 years and more
* Lung tumour of clinical staging I to IIIB receiving curative lung resection

Exclusion Criteria:

* Diagnosis of non small lung cancer invalidated by the histological findings of the operative sample
* psychological conditions, social support or geographical conditions not allowing the study follow up
* Pre operative chemotherapy or radiotherapy

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients aged 70 years and more with Non Small Cell lung Cancer.
Sampling Method: Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2009-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Post operative morbidity à 30-day | March 2014
  Post operative morbidity at 30-day :
  Post operative complications occurred during 30 days post surgery, evaluated with CTCAE V3.0. Complications grade 2.3.4 will be analyzed from day 1 up to day 30, collected at Day 1,Day 10, Day 30.
  A data collection is scheduled at Day 90 for delayed complications.
  Evaluation :
  preoperative at Day-30 up to Day 0, Postoperative at Day 10, day 30, Day 90, Day 360.

SECONDARY OUTCOMES:
Post operative mortality | March 2014
  Post operative mortality : mortality from Day 1 to Day 30 and survival at Day 360.
  Quality of life will be evaluated by :
  LCSS Spitzer index ADL,IADL.
Length of post operative hospital stay | March 2014
  Length of post operative hospital stay : hospitalization duration : intensive care, surgery department evaluated at Day 10 and post operative visit Day 30.
Length of intensive care unit stay | March 2014
  Length of intensive care unit stay evaluated at Day 10 (hospital release)and post operative visit at Day 30

CONTACTS AND LOCATIONS:
Overall Officials: LECAER HERVE, MD, Study Director — HOPITAL DE DRAGUIGNAN - SERVICE DE PNEUMOLOGIE; CHOUAID CHRISTOS, PR, Study Director — HOPITAL INTERCOMMUNAL DE CRETEIL SERVICE DE PNEUMOLOGIE; RAYNAUD Christine, MD, Principal Investigator — CENTRE HOSPITALIER D'ARGENTEUIL
Locations (25):
- France (25):
  - Centre Hospitalier D Argenteuil, Argenteuil, Val D'oise
  - Site 12, Aix-en-Provence
  - Centre Hospitalier Universitaire, Angers
  - Centre Hospitalier du Morvan, Brest
  - Centre François Baclesse, Caen
  - Centre Hospitalier René Dubos, Cergy-Pontoise
  - Site 30, Charleville-Mézières
  - Site 33, Créteil
  - Site 07, Draguignan
  - Site 32, Elbeuf
  - Site 04, Gap
  - Centre Hospitalier Les Oudairies, La Roche-sur-Yon
  - Site 41, Le Chesnay
  - Hospital du Cluzeau, Limoges
  - Centre Hospitalier Régional, Longjumeau
  - Site 06, Marseille
  - Site 42, Orléans
  - Hospital Saint Antoine, Paris
  - Site 19, Périgueux
  - Site 20, Rennes
  - Site 18, Rouen
  - Site 17, Rouen
  - Hôpital Yves Le Foll, Saint-Brieuc
  - Site 14, Toulon
  - Site 11, Villefranche-sur-Saône